CLINICAL TRIAL: NCT04721912
Title: Open-label Randomized Control Trial and Feasibility Study of Florjajen Digestion Probiotics to Reduce GBS Colonization in Pregnant Women by the Time of Birth.
Brief Title: Group B Streptococcus Response After Probiotic Exposure
Acronym: GRAPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Marquette University (Other)
Responsible Party: Principal Investigator, Katrina A. Nardini, Principle Investigator, CNM, WHNP-BC, MPH, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-396
Record Dates: First submitted 2020-12-07; First posted 2021-01-25 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Group B Strep Infection
Keywords: pregnancy; Group B Strep positive
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Intervention Model Description: Healthy pregnant participants will be randomly assigned to one of two groups (Probiotic vs No Probiotic (standard of care)). The Probiotic group will take one capsule daily and have the same study measures at the same times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care (No Intervention): Subjects in the control group will not receive any Probiotic capsules and will be advised to continue their routine prenatal self-care.
- Probiotic Dietary Supplement (Experimental): Participants in the intervention group will begin taking oral study Probiotic capsules once daily from time of enrollment/randomization at ≥ 36 weeks gestation until the time of birth. The research staff member will sequentially distribute the pre-labeled bottles of study capsules to the intervention group, one bottle of 30 Florajen Digestion probiotic capsules to women in the intervention group at the time of randomization.
  Interventions: Drug: Probiotic dietary supplement

INTERVENTIONS:
Drug: Probiotic dietary supplement — GBS positive patients, at ≥ 36 weeks gestation, will begin taking oral Florajen Digestion probiotic capsules once daily from time of enrollment/randomization at ≥ 36 weeks gestation until the time of birth.
  Other Names: Florajen Digestion™
  Arms: Probiotic Dietary Supplement

SUMMARY:
This is an open-label randomized control trial and feasibility study designed to determine the feasibility of a larger RCT in our setting that would examine prenatal probiotic use in Group B Strep (GBS) positive pregnant women at term. Investigators hope to address the question of whether prenatal oral probiotic use, taken by healthy low risk GBS positive women from approximately 37 weeks gestation until the time of birth, will reduce the number of women who test positive for GBS at the time of admission to Labor and Delivery (L&D).

DETAILED DESCRIPTION:
This is an open-label randomized control trial and feasibility study designed to determine the feasibility of a larger RCT in our setting that would examine prenatal probiotic use in Group B Strep (GBS) positive pregnant women at term. We hope to address the question of whether prenatal oral probiotic use, taken by healthy low risk GBS positive women from approximately 37 weeks gestation until the time of birth, will reduce the number of women who test positive for GBS at the time of admission to Labor and Delivery (L&D). In this study we aim to determine whether such a study is acceptable in our population, whether any adverse events are identified, and what barriers or confounding variables might exist to probiotic use at term. We will also look at whether probiotic use had any reported effect on maternal gastrointestinal (GI) symptoms.

ELIGIBILITY:
Inclusion Criteria:

• Healthy adult (≥ 18 years of age) pregnant women who are 36 - 37 6/7 weeks gestation at enrollment [calculated from the first day of Last Normal Menstrual Period (LNMP) and/or ultrasound (US)]

Group B Streptococcus Positive at 36 weeks gestation with:

* No obstetric complication requiring delivery prior to 39 weeks (hypertensive disorder diagnosed prior to enrollment, gestational diabetes, multiple gestation)
* No fetal complication (e.g., birth defect, intrauterine growth restriction)
* No medical complication (e.g., chronic hypertension, preexisting diabetes mellitus)
* Who do not currently ingest an over the counter probiotic supplement (not including yogurt)
* Who can both speak and read English or Spanish
* Pregnant women who regularly attend UNM prenatal clinics for their prenatal care ("regularly attend" will be defined as starting prenatal care prior to 20 weeks gestation and missing no more than one prenatal appointment during this pregnancy)
* No hypersensitivity reaction to β-lactam antibiotics

Exclusion Criteria:

* Those less than 18 years of age
* Non-pregnant women
* Later in pregnancy than 38 weeks gestation at enrollment [per LNMP and/or US]
* Those with an obstetric, fetal or medical complication of pregnancy
* Group B Streptococcus negative at 36 weeks gestation. Those ineligible for testing at 36 weeks gestation (history of GBS bacteriuria during the current pregnancy or have previously given birth to a GBS affected child.) We will not exclude those with bacteriuria other than GBS, and we will not exclude women who have taken an antibiotic during pregnancy, but we will track this as it is addressed in the Questionnaire for Women.
* Women who are currently ingesting an over the counter probiotic supplement (except for yogurt)
* Women who do not have electricity in the home.
* Women who are planning an elective repeat cesarean birth
* Women who do not speak and read English or Spanish
* Women with a history of missing one or more scheduled prenatal visit during this pregnancy
* Hypersensitivity reaction to β-lactam antibiotics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katrina Nardini, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Hospital, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Nardini K, Hanson L, Borders N, Singh M, Shields A, Trujillo VY, Lawton R, Malloy E. Open-Label Randomized Controlled Trial and Feasibility Study of an Oral Probiotic Intervention to Reduce Group B Streptococcus Colonization in Pregnant People by the Time of Birth. J Midwifery Womens Health. 2025 May-Jun;70(3):460-467. doi: 10.1111/jmwh.13765. Epub 2025 May 29. PMID 40442923

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Probiotic Dietary Supplement
Started | 34 | 34
Completed | 21 | 25
Not Completed | 13 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Probiotic Dietary Supplement | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Although 68 participants were randomized, 3 withdrew prior to obtaining age data and thus were not included in analysis.
  years
    number analyzed (Participants) | 33 | 32 | 65
    (all) | 28.8788 (5.40693) | 29.9688 (6.36261) | 29.42 (5.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 20 | 40
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 0 | 3 | 3
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Black or African American | 1 | 0 | 1
  Race: White | 21 | 21 | 42
  Race: More than one race | 2 | 1 | 3
  Race: Unknown or Not Reported | 10 | 9 | 19
Relationship Status [Count of Participants; unit: Participants]
  Single/widowed | 7 | 12 | 19
  Partnered/married | 24 | 18 | 42
  Missing | 3 | 4 | 7
Living Arrangements [Count of Participants; unit: Participants]
  Lives with others | 29 | 28 | 57
  Lives alone | 2 | 2 | 4
  Missing | 3 | 4 | 7
Education Level [Count of Participants; unit: Participants]
  HS/GED/some college | 10 | 10 | 20
  College | 12 | 13 | 25
  Graduate Degree | 9 | 7 | 16
  Missing | 3 | 4 | 7
Socio-economic status [Count of Participants; unit: Participants]
  <$40,000 | 7 | 7 | 14
  $40,000-99,999 | 8 | 12 | 20
  >$100,000 | 9 | 9 | 18
  Prefer not to answer | 7 | 0 | 7
  Missing | 3 | 6 | 9
Parity [Count of Participants; unit: Participants]
  Nulliparous | 13 | 11 | 24
  Multiparous | 20 | 20 | 40
  Missing | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: GBS Culture Result (Positive Versus Negative)
Description: Qualitative GBS colonization (positive versus negative)
Time Frame: T2 (admission to Labor and Delivery; 36 - 42 weeks gestational age)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Probiotic Dietary Supplement
Number analyzed (Participants) | 21 | 25
Participants
  Negative Qualitative GBS Colonization | 3 | 6
  Positive Qualitative GBS Colonization | 18 | 19

2. Secondary Outcome: Probiotic Pill Count to Measure Intervention Adherence
Description: Intervention adherence by pill count for probiotic participants
Time Frame: T3 (Postpartum day 0-14, up to 8 weeks from Baseline)
Population: Standard of Care participants did not receive probiotics and thus did not possess probiotic capsules to count and thus this analysis does not apply to this group.
Measure: Mean (Standard Deviation); unit: Average Florajen Digestion Pills
Arm/Group | Standard of Care | Probiotic Dietary Supplement
Number analyzed (Participants) | 0 | 25
Average Florajen Digestion Pills |  | 14 (7.87)

3. Secondary Outcome: Antepartum Gastrointestinal Symptom Assessment (AP-GI-SA) Score
Description: Maternal gastrointestinal (GI) symptoms based on AP-GI-SA score: lowest score 10, highest score 50 (high score means more symptoms = worse outcome)
Time Frame: Baseline T1 (36-37.6 weeks gestational age) and T3 (postpartum day 0-14; up to 8 weeks from baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care | Probiotic Dietary Supplement
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 15.6 (3.3) | 15.0 (3.3)
  Post-birth | 14.5 (4.8) | 13.5 (4.7)

4. Secondary Outcome: Number of Participants Who Report Adverse Events
Description: Maternal adverse events by organ system and severity.
Time Frame: T1 (baseline; 36.0-37.6 weeks gestational age) through T5 (6 weeks postpartum visit; up to 12 weeks and 6 days from baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Probiotic Dietary Supplement
Number analyzed (Participants) | 21 | 25
Participants | 0 | 0

5. Secondary Outcome: Number of Participants Who Report Adverse Events in Their Infant
Description: Infant adverse events by organ system and severity
Time Frame: T2 (admission to Labor and Delivery; 36 - 42 weeks gestational age) through T5 (6 weeks postpartum visit; up to 12 weeks and 6 days from baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Probiotic Dietary Supplement
Number analyzed (Participants) | 21 | 25
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: T1 (baseline; 36.0-37.6 weeks) through T5 (6 week postpartum visit; up to 12 weeks and 6 days from baseline)
Description: We did not find any reports of adverse events in our study participants.
Arm/Group | Standard of Care | Probiotic Dietary Supplement
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34

LIMITATIONS AND CAVEATS:
Participants and researchers were not masked to group assignment which may have led to unintended biases in responses and interpretation of questionnaires. Several IP samples were missed. The COVID-19 pandemic limited recruitment and may have prevented recruitment of those who would otherwise have participated. There were significant problems with laboratory processing of IP GBS swabs, resulting in 23 laboratory samples not being analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT04721912/Prot_SAP_000.pdf